CLINICAL TRIAL: NCT03917654
Title: Safety, Immunogenicity and Efficacy of Pfs230D1M-EPA/AS01 Vaccine, a Transmission Blocking Vaccine Against Plasmodium Falciparum, in an Age De-Escalation Trial of Children and a Family Compound Trial in Mali
Brief Title: Pfs230D1M-EPA/AS01 Vaccine, a Transmission Blocking Vaccine Against Plasmodium Falciparum, in an Age De-Escalation Trial of Children and a Family Compound Trial in Mali
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 999919086; 19-I-N086
Record Dates: First submitted 2019-04-16; First posted 2019-04-17 (Actual); Results first posted 2022-08-23 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2021-12

CONDITIONS: Malaria
Keywords: Randomized; Assays; Blood Smear; Antibody; Parasites
MeSH Terms: conditions — Malaria | interventions — Hepatitis A Vaccines; Vi polysaccharide vaccine, typhoid; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Arm 1a/3c (Experimental): Arm 1a (pilot) + Arm 3c (main) to receive 40ug of Pfs230D1M-EPA/AS01 on days 0, 28, 168; receipt of artemether/lumefantrine (AL) on day -7
  Interventions: Biological: Pfs230D1M-EPA/AS01; Biological: AVAXIM
- Arm 1b/3d (Active Comparator): Arm 1b (pilot) + Arm 3d (main) to receive HAVRIX (day 0), TYPHIM Vi (day 28), HAVRIX (day 168); receipt of AL on day -7
  Interventions: Biological: HAVRIX; Biological: Menactra
- Arm 2a/3a (Experimental): Arm 2a (pilot) + Arm 3a (main) to receive 40ug of Pfs230D1M-EPA/AS01 on days 0, 28, 168; receipt of AL on day -7 and 154
  Interventions: Biological: Pfs230D1M-EPA/AS01
- Arm 2b/3b (Active Comparator): Arm 2b (pilot) + Arm 3b (main) to receive HAVRIX (day 0), TYPHIM Vi (day 28), HAVRIX (day 168); receipt of AL on day -7 and 154
  Interventions: Biological: HAVRIX; Biological: Menactra
- Arm 3e (Experimental): Arm 3e (main) to receive 40microg of Pfs230D1M-EPA/AS01 on days 0, 28, 168; receipt of AL on day -7
  Interventions: Biological: Pfs230D1M-EPA/AS01
- Arm 3f (Active Comparator): Arm 3f (main) to receive HAVRIX (day 0), TYPHIM Vi (day 28), HAVRIX (day 168); receipt of AL on day -7
  Interventions: Biological: HAVRIX; Biological: TYPHIM Vi (Salmonella typhi vaccine); Biological: Menactra
- Arm 4a (No Intervention): Receipt of AL on day 154
- Arm 4b (No Intervention): Receipt of AL on day 154

INTERVENTIONS:
Biological: Pfs230D1M-EPA/AS01 — The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM phosphate-buffered saline (PBS) to a 2X dilution of the high dose (160 (Micro)g/mL in 0.5 mL volume) in cGMP compliance at Walter Reed Bioproduction facility in April 2016 and will be provided as a single use vial. AS01B adjuvant was manufactured for use in the SHINGRIX vaccine by GSK
  Arms: Arm 1a/3c; Arm 2a/3a; Arm 3e
Biological: HAVRIX — HAVRIX (Hepatitis A Vaccine; HAV) is produced by GSK and is a sterile suspension of inactivated virus for IM administration. The virus (strain HM175) is propagated in MRC-5 human diploid cells. HAVRIX is FDA approved for active immunization against disease caused by HAV for persons 12 months of age and older.
  Arms: Arm 1b/3d; Arm 2b/3b; Arm 3f
Biological: TYPHIM Vi (Salmonella typhi vaccine) — TYPHIM Vi (Typhoid Vi Polysaccharide Vaccine), produced by Sanofi Pasteur SA, for IM use, is a sterile solution containing the cell surface Vi polysaccharide extracted from Salmonella enterica serovar Typhi, S typhi Ty2 strain (inactivated, subunit vaccine). TYPHIM Vi vaccine is indicated for active immunization for the prevention of typhoid fever caused by S typhi and is FDA approved for use in persons 2 years of age or older
  Arms: Arm 3f
Biological: Menactra — Menactra (Sanofi Pasteur) is a sterile, intramuscularly administered vaccine that contains Neisseria meningitidis serogroup A, C, Y, and W-135 capsular polysaccharide antigens individually conjugated to diphtheria toxoid protein. No preservative or adjuvant is added during the manufacturing process. Menactra is FDA approved for active immunization to prevent invasive meningococcal disease caused by Neisseria meningitidis serogroups A, C, Y, and W-135 (but does not protect against serotype B) for use in individuals 9 months through 55 years of age.
  Arms: Arm 1b/3d; Arm 2b/3b; Arm 3f
Biological: AVAXIM — AVAXIM - Pediatric [Hepatitis A Vaccine Inactivated] is a sterile, whitish, cloudy suspension. The active ingredient is a purified and formaldehyde-inactivated hepatitis A virus (HAV) obtained from the GBM strain, cultured on MRC-5 human diploid cells. HAV is adsorbed onto aluminum.
  Arms: Arm 1a/3c

SUMMARY:
Background:

Malaria affects many people in Mali and other parts of Africa. It is spread by mosquito bites. Malaria can make people sick or can lead to death. Scientists want to learn if a vaccine can stop it from spreading to other people.

Objective:

To test how well an experimental malaria vaccine works to decrease malaria infections.

Eligibility:

Healthy people ages 5 and older who live in Doneguebougou, Mali, and surrounding areas

Design:

Participants will be screened with:

Medical history

Physical exam

Blood, urine, and heart tests

EKG

Participants will be randomly assigned to get either the experimental vaccine or an approved vaccine. They will not know which they are getting.

Participants will have a visit about a week before their first vaccine. They will take a medicine that kills malaria. They will take it at the clinic the next 2 days. Participants ages 5-8 will take the drug again 2 weeks before their third vaccine.

Participants get the vaccine through a needle in the arm. They will have visits 1, 3, 7, and 14 days after. They will have blood tests or finger pricks.

Participants will get another vaccine 1 and 6 months later.

Participants will have blood tests once a month. At these visits they may also have urines tests or mosquito feeds. For the feeds a cup full of mosquitoes will be placed on arms or legs for 15-20 minutes.

Participants will have visits twice a month for 4 months after their last vaccine.

DETAILED DESCRIPTION:
A vaccine to interrupt malaria transmission (VIMT), targeting disruption of both human and mosquito transmission, would be a valuable tool for local elimination or eradication of this disease. One strategy to design a VIMT is using components that block transmission of malaria to mosquitoes, such as Pfs230. Pfs230, a surface antigen of intracellular gametocytes, as well as extracellular gametes and zygotes in the mosquito stage of Plasmodium falciparum, is currently the leading candidate in clinical trials for a malaria transmission-blocking vaccine (TBV). Recombinant Pfs230D1M has been conjugated to a recombinant Pseudomonas aeruginosa ExoProtein A (EPA) and adjuvanted with AS01. When formulated in AS01, results from a recent first-in-human trial demonstrated that Pfs230-EPA induces functional transmission-reducing, and in a significant proportion of vaccinees, transmission-blocking serum activity that can be measured for months, the vaccine is well-tolerated and safe in adults, and our recent natural history data clearly indicate that children play a disproportionate role in malaria transmission. The next step in the development of Pfs230D1M-EPA as a TBV is therefore to conduct an age de-escalation trial to ensure that the vaccine is safe to administer to children and then to conduct a community clinical trial to assess efficacy in family groups.

This Phase 2 study will first determine safety and tolerability of Pfs230D1M-EPA/AS01 in healthy Malian children of decreasing ages: 9-18 years old, followed by 5-8 years old. A total of 60 subjects will be enrolled in Doneguebougou, Mali, West Africa. Children will be recruited from compounds/family that have agreed to participate in the main phase of the study and will enroll in a staggered manner to receive either Pfs230D1M-EPA/AS01 vaccine or comparator as assigned by their compound block randomization. Prior to receipt of vaccination #1, all subjects will receive a full treatment course of artemether/lumefantrine (AL). Safety and tolerability will be monitored and reported as local and systemic adverse events (AEs) and serious adverse events (SAEs) and reviewed by DSMB, sponsor, medical monitors, and study team prior to proceeding with enrollment of the main phase.

If there are no safety concerns, in a staggered manner, the main phase will begin enrollment of approximately 137 compounds/vaccine units (about 1500 vaccinees + about 400 under 5 years of age for parasite surveillance). Children enrolled during the pilot safety phase will join their main phase compounds/family for vaccination #3. Prior to receipt of first vaccination, all subjects will receive a full treatment course of AL. All vaccinated subjects will be monitored for safety and tolerability. Immunogenicity outcomes will be antibody responses as measured by enzyme-linked immunosorbent assay (ELISA) against recombinant Pfs230D1M. Functional activity of the induced antibodies will be assessed by standard membrane feeding assays in select samples. Vaccine activity will be measured in children 9-18 years of age who will undergo direct skin feeds (DSF) starting 2 weeks post vaccination #3 for a total of 8 DSFs.

Prior to scheduled last vaccination in members of the compound/family, children 1-4 years of age and vaccinated children 5-8 years of age will receive a full treatment course of AL prior to the expected start of the transmission season and will then be followed every 2 weeks by blood smear (BS) along with all vaccinated children. Children 9-18 years of age will also be assessed for vaccine efficacy, but as a separate analysis from those 1-8 years of age.

In Year 2, those who received vaccination during Year 1 (5 years of age and older at enrollment), if eligible and still on study, will receive a single fourth vaccination per their vaccine unit (VU) blinded arm assignment. No new individuals will be enrolled. Again, children 1-4 years of age and vaccinated children 5-8 years of age will receive a full treatment course of AL prior to the expected start of the transmission season and will then be followed every 2 weeks by BS along with all vaccinated children. Children 9-18 years of age will also be assessed for vaccine efficacy against parasitemia, but as a separate analysis from those 1-8 years of age. Immunogenicity outcomes will be antibody responses as measured by ELISA against recombinant Pfs230D1M. Functional activity of the induced antibodies will be assessed by standard membrane feeding assays in select samples. Vaccine activity will be measured in children 9-18 years of age who will undergo DSF starting 2 weeks post vaccination #4 for a total of 10 DSFs.

ELIGIBILITY:
* INCLUSION CRITERIA FOR GROUPS 1,2,3:

All of the following criteria must be fulfilled for a volunteer to participate in this trial:

1. Meets age requirements for Arm currently being enrolled.
2. Available for the duration of the trial.
3. Family compound known resident or long-term resident (more than 1 year) of Doneguebougou, Mali or surrounding villages.
4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
5. In good general health and without clinically significant medical history in the opinion of the investigator.
6. Females of childbearing potential must be willing to use reliable contraception from 21 days prior to Study Day 0 and until 1 month after the last vaccination.

   * A reliable method of birth control includes one of the following:

<!-- -->

1. Confirmed pharmacologic contraceptives (parenteral) delivery;
2. Intrauterine or implantable device

EXCEPTIONS to required pregnancy prevention includes the following:

1. Postmenopausal state: defined as no menses for 12 months without an alternative medical cause
2. Surgical sterilization
3. Unmarried AND not sexually active AND menstruating OR not menstruating females 12-17 years of age
4. NOTE: if a female of childbearing potential s status changes during the course of vaccination through 1 month post vaccination (e.g. they become >=18 years of age, married, or sexually active), the female will be required to start reliable contraception

7. Willing to have blood samples stored for future research.

INCLUSION CRITERIA FOR GROUP 4:

All of the following criteria must be fulfilled for a volunteer to participate in this trial:

1. Meets age requirements for Arm currently being enrolled.
2. Available for the duration of the trial.
3. Family compound known resident or long-term resident (more than 1 year) of Doneguebougou, Mali or surrounding villages.
4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
5. In good general health and without clinically significant medical history in the opinion of the investigator.
6. Willing to have blood samples stored for future research.

Inclusion Criteria for Groups 1, 2, 3, (Year 2)

All of the following criteria must be fulfilled for a volunteer to continue to participate in this trial:

1. Previously enrolled in the study and has received at least 1 vaccination. 2. Available for the duration of the trial.

3. In good general health and without clinically significant medical history in the opinion of the investigator.

4. Females of childbearing potential must be willing to use reliable contraception from 21 days prior to scheduled vaccine dose #4 and until 1 month after the 4th vaccination.

-A reliable method of birth control includes one of the following:

1. Confirmed pharmacologic contraceptives (parenteral) delivery;
2. Intrauterine or implantable device

EXCEPTIONS to required pregnancy prevention includes the following:

1. Postmenopausal state: defined as no menses for 12 months without an alternative medical cause
2. Surgical sterilization
3. Unmarried AND not sexually active AND menstruatingOR not menstruating females 12-17 years of age
4. NOTE: if a female of childbearing potential s status changes during the course of vaccination through 1 month post vaccination (e.g. they become greater than or equal to 18 years of age, married, or sexually active), the female will be required to start reliable contraception
5. Willing to have blood samples stored for future research.

Inclusion Criteria for Group 4 (Year 2):

All of the following criteria must be fulfilled for a volunteer to continue to participate in this trial:

1. Previously enrolled in the study
2. Available for the duration of the trial.
3. In good general health and without clinically significant medical history in the opinion of the investigator.
4. Willing to have blood samples stored for future research.

EXCLUSION CRITERIA FOR GROUPS 1, 2, 3:

An individual will be excluded from participating in this trial if any one of the following criteria is fulfilled:

1. Pregnant, as determined by a positive urine or serum beta human choriogonadotropin (beta-hCG) test (if female).

   NOTE: Pregnancy is also a criterion for discontinuation of any further vaccine dosing
2. Menstruating females 11 years of age and younger. (In order to avoid cultural implications of further assessing pregnancy potential i.e. sexual activity in this age group.)
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and comply with the study protocol at a level appropriate for the subject s age.
4. Hemoglobin, white blood cell (WBC), absolute neutrophil count, or platelet levels outside the local laboratory defined limits of normal. (Subjects may be included at the investigator s discretion for not clinically significant values outside of normal range and <= Grade 2.)
5. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory defined upper limit of normal. (Subjects may be included at the investigator s discretion for not clinically significant values outside of normal range and <= Grade 2.)
6. Infected with HIV
7. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
8. Clinically significant prolonged QTc (>450 milliseconds) on screening EKG
9. History of receiving any investigational product within the past 30 days.
10. Current or planned participation in an investigational vaccine study until the last required protocol visit.
11. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
12. History of a severe allergic reaction or anaphylaxis.
13. Known:

    * Severe asthma, defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years.
    * Autoimmune or antibody-mediated disease including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sj(SqrRoot)(Delta)gren s syndrome, or autoimmune thrombocytopenia.
    * Immunodeficiency syndrome.
    * Seizure disorder (exception: history of simple febrile seizures)
    * Asplenia or functional asplenia.
    * Use of chronic (>=14 days) oral or intravenous (IV) corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of Study Day 0.
    * Allergy to latex or neomycin
    * Adverse reaction to hepatitis A and/or typhoid and/or meningococcal vaccine in the past
    * Adverse reaction to artemether/lumefantrine in the past
14. Receipt of:

    -Live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks to enrollment.
    * Immunoglobulins and/or blood products within the past 6 months.
    * Investigational malaria vaccine in the last 2 years.
15. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.

Co-enrollment guidelines: Co-enrollment in other trials is restricted, other than enrollment on observational studies. Consideration for co-enrollment in trials evaluating the use of a licensed medication will require the approval of the PI. Study staff should be notified of co-enrollment on any other protocol as it may require the approval of the investigator.

Exclusion Criteria for Group 4:

An individual will be excluded from participating in this trial if any one of the following criteria is fulfilled:

1. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and comply with the study protocol at a level appropriate for the subject s age.
2. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
3. Clinically significant prolonged QTc (by sex/age) on screening EKG
4. History of adverse reactions to artemether/lumefantrine in the past
5. History of receiving any investigational product within the past 30 days.
6. Current or planned participation in an investigational vaccine study until the last required protocol visit.
7. Receipt of:

   -Investigational malaria vaccine in the last 2 years.
8. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.

Exclusion Criteria for Groups 1, 2, 3 (Year 2):

An individual will be excluded from participating in this trial if any one of the following criteria is fulfilled:

1. Pregnant, as determined by a positive urine or serum beta human choriogonadotropin (beta-hCG) test (if female).

   NOTE: Pregnancy is also a criterion for discontinuation of any further vaccine dosing
2. Menstruating females 11 years of age and younger. (In order to avoid cultural implications of further assessing pregnancy potential i.e. sexual activity in this age group.)
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and comply with the study protocol at a level appropriate for the subject s age.
4. Hemoglobin, white blood cell (WBC), absolute neutrophil count, or platelet levels outside the local laboratory defined limits of normal. (Subjects may be included at the investigator s discretion for not clinically significant values outside of normal range and less than or equal to Grade 2.)
5. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory defined upper limit of normal. (Subjects may be included at the investigator s discretion for not clinically significant values outside of normal range and less than or equal to Grade 2.)
6. Infected with HIV
7. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
8. History of receiving any investigational product within the past 30 days.
9. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
10. History of a severe allergic reaction or anaphylaxis.
11. Known:

    -Severe asthma, defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years.

    -Autoimmune or antibody-mediated disease including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren s syndrome, or autoimmune thrombocytopenia.
    * Immunodeficiency syndrome.
    * Seizure disorder (exception: history of simple febrile seizures)
    * Asplenia or functional asplenia.
    * Use of chronic (greater than or equal to 14 days) oral or intravenous (IV) corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of Study Day 0.
    * Allergy to latex or neomycin
    * Adverse reaction to hepatitis A and/or typhoid and/or meningococcal vaccine in the past
    * Adverse reaction to artemether/lumefantrine in the past
12. Receipt of:

    * Live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks to enrollment.
    * Immunoglobulins and/or blood products within the past 6 months.
13. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.

Exclusion Criteria for Group 4 (Year 2):

An individual will be excluded from participating in this trial if any one of the following criteria is fulfilled:

1. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and comply with the study protocol at a level appropriate for the subject s age.

2. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.

3. History of adverse reactions to artemether/lumefantrine in the past

4. History of receiving any investigational product within the past 30 days.

5. Current or planned participation in an investigational vaccine study until the last required protocol visit.

6. Receipt of:

* Investigational malaria vaccine in the last 2 years.

  7. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1301 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Mrtc/Usttb, Bamako, Mali

REFERENCES:
- [Background] MacDonald NJ, Nguyen V, Shimp R, Reiter K, Herrera R, Burkhardt M, Muratova O, Kumar K, Aebig J, Rausch K, Lambert L, Dawson N, Sattabongkot J, Ambroggio X, Duffy PE, Wu Y, Narum DL. Structural and Immunological Characterization of Recombinant 6-Cysteine Domains of the Plasmodium falciparum Sexual Stage Protein Pfs230. J Biol Chem. 2016 Sep 16;291(38):19913-22. doi: 10.1074/jbc.M116.732305. Epub 2016 Jul 18. PMID 27432885
- [Background] Tachibana M, Wu Y, Iriko H, Muratova O, MacDonald NJ, Sattabongkot J, Takeo S, Otsuki H, Torii M, Tsuboi T. N-terminal prodomain of Pfs230 synthesized using a cell-free system is sufficient to induce complement-dependent malaria transmission-blocking activity. Clin Vaccine Immunol. 2011 Aug;18(8):1343-50. doi: 10.1128/CVI.05104-11. Epub 2011 Jun 29. PMID 21715579
- [Background] Farrance CE, Rhee A, Jones RM, Musiychuk K, Shamloul M, Sharma S, Mett V, Chichester JA, Streatfield SJ, Roeffen W, van de Vegte-Bolmer M, Sauerwein RW, Tsuboi T, Muratova OV, Wu Y, Yusibov V. A plant-produced Pfs230 vaccine candidate blocks transmission of Plasmodium falciparum. Clin Vaccine Immunol. 2011 Aug;18(8):1351-7. doi: 10.1128/CVI.05105-11. Epub 2011 Jun 29. PMID 21715576
- [Derived] Cao Y, da Silva Araujo M, Lorang CG, Dos Santos NAC, Tripathi A, Vinetz J, Kumar N. Distinct immunogenicity outcomes of DNA vaccines encoding malaria transmission-blocking vaccine target antigens Pfs230D1M and Pvs230D1. Vaccine. 2025 Feb 15;47:126696. doi: 10.1016/j.vaccine.2024.126696. Epub 2025 Jan 8. PMID 39787798

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1a: Pilot/safety: Dosing interval on days: 0, 28, 126, 448
  Participants received 4 doses of 40 μg of Pfs230D1M-EPA/AS01 administered via intramuscular (IM) injection on days: 0, 28, 126, 448; receipt of artemether/lumefantrine (AL) on day -7
- Arm 1b: Pilot/safety: Dosing interval on days: 0, 28, 126, 448
  Participants received 4 doses administered via intramuscular (IM) injection on days 0, 448 to receive HAVRIX; day 28 to receove TYPHIM Vi; and day 126 to receive Menactra; receipt of AL on day -7
- Arm 2a: Pilot/safety: Dosing interval on days: 0, 28, 126, 448
  Participants received 4 doses administered via intramuscular (IM) injection on days 0, 28, 126, 448 to receive 40 μg of Pfs230D1M-EPA/AS01; receipt of AL on day -7,112, 441
- Arm 2b: Pilot/safety: Dosing interval on days: 0, 28, 126, 448
  Participants received 4 doses administered via intramuscular (IM) injection on days 0, 448 to receive HAVRIX; day 126 to receive Menactra; receipt of AL on day -7,112, 441
- Arm 3a: Safety/efficacy: Dosing interval on days 0, 28, 56, 392
  Participants received 4 doses administered via intramuscular (IM) injection on days 0, 28, 56, 392 to receive 40 μg of Pfs230D1M-EPA/AS01; receipt of AL on day -7, 42, 385
- Arm 3b: Safety/efficacy: Dosing interval on days 0, 28, 56, 392
  Participants received 4 doses administered via intramuscular (IM) injection on days 0, 392 to receive HAVRIX; day 28 TYPHIM Vi; day 56 to receive Menactra; receipt of AL on day -7, 42, 385
- Arm 3c; Arm 3e: Safety/efficacy: Dosing interval on days 0, 28, 56, 392
  Participants received 4 doses administered via intramuscular (IM) injection on days 0, 28, 56, 392 to receive 40 μg of Pfs230D1M-EPA/AS01; receipt of AL on day -7
- Arm 3d; Arm 3f: Safety/efficacy: Dosing interval on days 0, 28, 56, 392
  Participants received 4 doses administered via intramuscular (IM) injection on days 0, 392 to receive HAVRIX; day 28 TYPHIM Vi; day 56 to receive Menactra; receipt of AL on day -7
- Arm 4a; Arm 4b: AL treatment only; no vaccination
  Participants received AL on day -14, 385
Period: Year 1
Arm/Group | Arm 1a | Arm 1b | Arm 2a | Arm 2b | Arm 3a | Arm 3b | Arm 3c | Arm 3d | Arm 3e | Arm 3f | Arm 4a | Arm 4b
Started | 15 | 15 | 15 | 15 | 99 | 87 | 192 | 177 | 227 | 267 | 97 | 95
Completed | 14 | 13 | 13 | 15 | 94 | 82 | 173 | 162 | 218 | 257 | 92 | 87
Not Completed | 1 | 2 | 2 | 0 | 5 | 5 | 19 | 15 | 9 | 10 | 5 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 2 | 5 | 3 | 1 | 0
Not completed — Travel | 0 | 1 | 1 | 0 | 4 | 4 | 10 | 8 | 2 | 5 | 3 | 3
Not completed — Subject moved away from site | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 3
Not completed — Spouse/Family member request | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Missed visits | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Period: Year 2
Arm/Group | Arm 1a | Arm 1b | Arm 2a | Arm 2b | Arm 3a | Arm 3b | Arm 3c | Arm 3d | Arm 3e | Arm 3f | Arm 4a | Arm 4b
Started (Year 2 participants did not equal Year 1 participants for each arm, due to a number of participants electing not to rescreen for Year 2.) | 13 | 10 | 13 | 14 | 86 | 77 | 152 | 147 | 199 | 238 | 90 | 87
Did Not Rescreen | 1 | 3 | 0 | 1 | 8 | 5 | 21 | 15 | 19 | 19 | 2 | 0
Completed | 10 | 9 | 13 | 14 | 82 | 75 | 138 | 139 | 185 | 226 | 89 | 83
Not Completed | 3 | 1 | 0 | 0 | 4 | 2 | 14 | 8 | 14 | 12 | 1 | 4
Not completed — Travel | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1
Not completed — Married | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Subject moved away from site | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 2 | 0 | 1
Not completed — Year 2 Screening failure | 0 | 1 | 0 | 0 | 2 | 0 | 4 | 3 | 10 | 2 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 5 | 0 | 0
Not completed — Spouse/family member request | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1a | Arm 1b | Arm 2a | Arm 2b | Arm 3a | Arm 3b | Arm 3c | Arm 3d | Arm 3e | Arm 3f | Arm 4a | Arm 4b | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 99 | 87 | 192 | 177 | 227 | 267 | 97 | 95 | 1301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 15 | 15 | 99 | 87 | 178 | 167 | 0 | 0 | 97 | 95 | 783
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 10 | 208 | 249 | 0 | 0 | 481
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 18 | 0 | 0 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 5 | 6 | 50 | 43 | 84 | 91 | 126 | 147 | 44 | 43 | 653
  Male | 9 | 7 | 10 | 9 | 49 | 44 | 108 | 86 | 101 | 120 | 53 | 52 | 648
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Bambara | 9 | 11 | 6 | 2 | 51 | 34 | 84 | 51 | 115 | 139 | 41 | 32 | 575
  Sarakole | 6 | 3 | 8 | 11 | 45 | 51 | 93 | 121 | 98 | 122 | 45 | 58 | 661
  Peulh | 0 | 1 | 1 | 1 | 2 | 1 | 12 | 0 | 8 | 4 | 5 | 3 | 38
  Other | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 2 | 0 | 2 | 10
  Malinke | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 6 | 0 | 5 | 0 | 15
  Bozo | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Sonrhai | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Mali | 15 | 15 | 15 | 15 | 99 | 87 | 192 | 177 | 227 | 267 | 97 | 95 | 1301

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local and Systemic Adverse Events in Years 1 and 2
Description: Number of participants with local and systemic adverse events (AEs) graded by severity occurring within 7 days after each vaccine
Time Frame: Within 7 days after each vaccination at days, 0, 28, 126, 448 (for arms 1a, 1b, 2a, 2b), days 0, 28, 56, 392 (for arms 3a, 3b, 3c, 3d, 3e, 3f), days -14 and 385 (for arms 4a, 4b) and year 2 (for all arms)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1a | Arm 1b | Arm 2a | Arm 2b | Arm 3a | Arm 3b | Arm 3c | Arm 3d | Arm 3e | Arm 3f | Arm 4a | Arm 4b
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 99 | 87 | 192 | 177 | 227 | 267 | 97 | 95
Participants | 15 | 14 | 15 | 15 | 96 | 85 | 187 | 172 | 224 | 260 | 89 | 85

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm 1a | Arm 1b | Arm 2a | Arm 2b | Arm 3a | Arm 3b | Arm 3c | Arm 3d | Arm 3e | Arm 3f | Arm 4a | Arm 4b
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/99 | 1/87 | 0/192 | 0/177 | 2/227 | 5/267 | 0/97 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 1/99 | 1/87 | 0/192 | 2/177 | 2/227 | 7/267 | 0/97 | 1/95
Other Adverse Events (participants affected / at risk) | 15/15 | 14/15 | 15/15 | 15/15 | 95/99 | 84/87 | 187/192 | 170/177 | 222/227 | 253/267 | 89/97 | 84/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1a (N=15) | Arm 1b (N=15) | Arm 2a (N=15) | Arm 2b (N=15) | Arm 3a (N=99) | Arm 3b (N=87) | Arm 3c (N=192) | Arm 3d (N=177) | Arm 3e (N=227) | Arm 3f (N=267) | Arm 4a (N=97) | Arm 4b (N=95)
Bacterial Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Blood Creatinine Increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Drowning (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
ESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Pancreatic carcinoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Prostate adenoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Struck by lightning (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1a (N=15) | Arm 1b (N=15) | Arm 2a (N=15) | Arm 2b (N=15) | Arm 3a (N=99) | Arm 3b (N=87) | Arm 3c (N=192) | Arm 3d (N=177) | Arm 3e (N=227) | Arm 3f (N=267) | Arm 4a (N=97) | Arm 4b (N=95)
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (3) | 2 (4) | 15 (18) | 19 (25) | 24 (26) | 24 (30) | 8 (8) | 16 (17) | 8 (9) | 6 (6)
Abdominal Pain Upper (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 2 (2) | 3 (3) | 0 | 0
Abscess (Infections and infestations) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 1 (1) | 1 (1) | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 (3) | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 1 (2) | 0 | 0 | 0 | 5 (5) | 5 (5) | 6 (7) | 3 (3) | 8 (12) | 9 (9) | 0 | 0
Arteritis (Vascular disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 (8) | 9 (9) | 0 | 0
Arthropod sting (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
Asthenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (3) | 7 (7) | 8 (8) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 4 (5) | 6 (6) | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Blood creatinine inreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 12 (15) | 22 (28) | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 9 (10) | 13 (13) | 13 (13) | 10 (10) | 21 (24) | 14 (14) | 9 (10) | 14 (19)
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Chills (Nervous system disorders) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 4 (6) | 5 (5) | 9 (9) | 13 (13) | 0 | 0
Circumcision (Skin and subcutaneous tissue disorders) | 0 (0) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 (0) | 0 | 0 | 0 | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 | 0 | 0 | 4 (4) | 1 (1) | 2 (2) | 0 | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 | 1 (1) | 3 (3) | 6 (6) | 4 (4) | 17 (20) | 6 (6) | 6 (6) | 14 (15) | 6 (6) | 4 (4)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 2 (2) | 0 | 0
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 3 (3) | 4 (4) | 18 (20) | 20 (22) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 5 (7) | 7 (8) | 12 (14) | 14 (14) | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 4 (4) | 1 (1) | 14 (15) | 16 (19) | 0 | 0
Dysentery (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 1 (1) | 1 (1) | 0 | 2 (2) | 9 (9) | 14 (14) | 2 (2) | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 1 (1) | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 (3) | 0 | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Erysipelas (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 13 (13) | 4 (4) | 0 | 0
Food poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 2 (2) | 0 | 2 (2) | 0 | 1 (1)
Forearm fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Foreign body in ear (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Fungal skin infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Furuncle (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 3 (3) | 3 (3) | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 3 (3) | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 3 (3) | 0 | 8 (8) | 9 (11) | 10 (10) | 13 (14) | 18 (20) | 22 (25) | 12 (13) | 10 (11)
Genital infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 5 (5) | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 8 (15) | 4 (6) | 7 (7) | 0 | 24 (29) | 6 (9) | 77 (117) | 46 (69) | 118 (182) | 100 (161) | 4 (4) | 0
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 (3) | 3 (5) | 5 (7) | 3 (3) | 6 (9) | 3 (3) | 0 | 0
Hordeolum (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Infection parasitic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Inflammation (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Injection site edema (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Injection site induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
Injection site movement impairment (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Injection site pain (Musculoskeletal and connective tissue disorders) | 15 (37) | 11 (21) | 15 (31) | 12 (19) | 80 (148) | 46 (74) | 148 (247) | 78 (105) | 152 (245) | 85 (106) | 0 | 0
Injection site pruritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 3 (3) | 0 | 0
Injection site swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Joint dislocation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Layrngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 | 0 | 0 | 0 | 3 (3) | 5 (6) | 3 (5) | 6 (7) | 3 (3) | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 | 1 (1) | 1 (1) | 6 (6) | 15 (22) | 20 (25) | 28 (50) | 40 (61) | 0 | 0
Ligament sprain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 | 0
Lip swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 13 (31) | 11 (21) | 10 (26) | 10 (16) | 70 (155) | 61 (128) | 148 (316) | 120 (241) | 104 (149) | 137 (184) | 48 (81) | 46 (69)
Malnutrition (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Mastitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 3 (3) | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 (4) | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 17 (18) | 16 (22) | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 16 (18) | 11 (11) | 12 (12) | 8 (8) | 13 (15) | 11 (11) | 16 (19) | 8 (9)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 5 (5) | 6 (7) | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 (7) | 2 (2) | 2 (2) | 3 (5) | 4 (5) | 11 (12) | 20 (33) | 33 (41) | 38 (59) | 53 (84) | 0 | 0
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 0 | 0 | 0 | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 0 | 0
Otitis media (Ear and labyrinth disorders) | 0 (0) | 0 | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 | 3 (3)
Paronychia (Infections and infestations) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1) | 0
Parotitis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Pharyngitis (Gastrointestinal disorders) | 4 (5) | 1 (1) | 7 (9) | 7 (14) | 30 (43) | 29 (38) | 29 (35) | 36 (50) | 24 (26) | 20 (23) | 23 (29) | 25 (29)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 (3) | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0
Pyoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 2 (2) | 0 | 1 (1) | 0 | 0 | 0
Pyrexia (General disorders) | 2 (2) | 1 (1) | 7 (9) | 2 (2) | 29 (34) | 11 (13) | 36 (44) | 8 (10) | 34 (37) | 19 (19) | 16 (17) | 5 (5)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 5 (8) | 8 (15) | 6 (13) | 57 (93) | 44 (76) | 100 (162) | 96 (149) | 103 (157) | 136 (211) | 56 (79) | 60 (96)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 | 0
Sciatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 4 (4) | 0 (0) | 0 | 0
Sinobronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 2 (2) | 0 | 10 (10) | 3 (4) | 7 (8) | 10 (11) | 9 (10) | 14 (14) | 7 (8) | 4 (6)
Snake bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1) | 0 | 0
Systolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 (3) | 1 (1) | 0 | 0
Tachycardia (Cardiac disorders) | 3 (3) | 0 | 0 | 0 | 1 (2) | 3 (4) | 0 | 0 | 0 | 0 | 4 (5) | 2 (3)
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 | 0 | 0 | 6 (7) | 4 (4) | 8 (8) | 5 (6) | 6 (8) | 9 (16) | 0 | 0
Tonsilitis (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 | 3 (3) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Typhoid fever (Infections and infestations) | 0 | 0 | 0 | 0 | 3 (3) | 0 | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 0 | 0 | 2 (2) | 3 (3) | 2 (2) | 3 (4) | 2 (2) | 2 (2) | 5 (5) | 0 | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 4 (4) | 6 (6) | 2 | 1 (1)
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 (3) | 0 | 4 (4) | 3 (3) | 6 (6) | 2 (2) | 7 (7) | 6 (6) | 3 (3) | 5 (5)
Wound (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 (1) | 1 (1) | 4 (5) | 6 (6) | 5 (5) | 9 (10) | 5 (5) | 5 (5) | 0 (0) | 3 (3)
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 3 (3) | 1 (1) | 5 (5) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT03917654/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT03917654/ICF_001.pdf